CLINICAL TRIAL: NCT00676871
Title: A Phase 1/2, Open-Label, Single-Arm, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Antitumor Activity of Continuous Intravenous Infusion of the Bispecific T-Cell Engager MEDI-538 In Adults With B-Cell Chronic Lymphocytic Leukemia(CLL)Who Have Residual Disease Following Previous Therapy for CLL
Brief Title: A Study to Evaluate the Safety, Tolerability, and Antitumor Activity of Continuous Intravenous Infusion of MEDI-538 in Adults With B-Cell Chronic Lymphocytic Leukemia (CLL)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Replacing this trial with a new trial.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Karen Kaucic, MD, MedImmune
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP155
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Experimental): MEDI-538
  Interventions: Drug: MEDI-538
- 2 (Experimental): MEDI-538
  Interventions: Drug: MEDI-538
- 3 (Experimental): MEDI-538
  Interventions: Drug: MEDI-538
- 4 (Experimental): MEDI-538
  Interventions: Drug: MEDI-538
- 5 (Experimental): MEDI-538
  Interventions: Drug: MEDI-538
- 6 (Experimental): MEDI-538
  Interventions: Drug: MEDI-538
- 7 (Experimental): MEDI-538
  Interventions: Drug: MEDI-538

INTERVENTIONS:
Drug: MEDI-538 — Dose one of MEDI 538 as a continuous IV infusion - dose level is 5 mg/m2/24h (Phase 1)
  Arms: 1
Drug: MEDI-538 — Dose two of MEDI 538 as a continuous IV infusion - dose level is 10 mg/m2/24h (Phase 1)
  Arms: 2
Drug: MEDI-538 — Dose three of MEDI 538 as a continuous IV infusion-dose level is 15mg/m2/24h (Phase 1)
  Arms: 3
Drug: MEDI-538 — Dose four of MEDI 538 as a continuous IV infusion - dose level is 30 mg/m2/24h(Phase 1)
  Arms: 4
Drug: MEDI-538 — Dose five of MEDI 538 as a continuous IV infusion - dose level is 45 mg/m2/24h (Phase 1)
  Arms: 5
Drug: MEDI-538 — Dose six of MEDI 538 as a continuous IV infusion - dose level is 60 mg/m2/24h (Phase 1)
  Arms: 6
Drug: MEDI-538 — Phase 2 part of the study, 20 to 60 patients will be treated with MEDI 538 as a continuous IV infusion through a central line catheter. The dose of MEDI-538 will be determined in the Phase 1 part of the study.
  Arms: 7

SUMMARY:
Phase 1:

* Evaluate the safety and tolerability of MEDI-538 given by escalated doses with continuous IV infusion for 4 weeks in adult patients with CLL.
* Determine the maximum tolerated dose (MTD) of MEDI-538 administered by continuous IV infusion for 4 weeks in this patient population
* Describe the pharmacokinetics (PK) of MEDI-538
* Describe the immunogenicity (IM) of MEDI-538
* Determine the overall response, which is defined as follows: (1) conversion from PD/SD to PR/nPR/CR or conversion from PR to nPR/CR using standard NCI-WG criteria; or (2) conversion from MRD positivity to MRD negativity using 4-color flow cytometry; and
* Describe any antitumor activity (ie, time to response and duration of response) of MEDI-538 in this patient population.

Phase 2:

* To determine the overall response in adult patients with CLL who have residual disease following previous therapy for CLL.
* Describe the safety,PK,and IM of MEDI-538
* Determine the time to MRD relapse
* Determine the antitumor activity (ie, time to response, duration of response,and time to progression [TTP])of MEDI-538 in this patient population.

DETAILED DESCRIPTION:
Phase 1:

* Evaluate the safety and tolerability of MEDI-538 at doses of 5, 10, 15, 30, 45, or 60 mg/m2/24h by continuous IV infusion for 4 weeks in adult patients with CLL who have measurable disease following previous therapy for CLL. Patients with measurable disease include patients who demonstrated PD, SD, or PR following previous therapy for CLL; and
* Determine the maximum tolerated dose (MTD) of MEDI-538 administered by continuous IV infusion for 4 weeks in this patient population;
* Describe the pharmacokinetics (PK) of MEDI-538
* Describe the immunogenicity (IM) of MEDI-538
* Determine the overall response, which is defined as follows: (1) conversion from PD/SD to PR/nPR/CR or conversion from PR to nPR/CR using standard NCI-WG criteria; or (2) conversion from MRD positivity to MRD negativity using 4-color flow cytometry; and
* Describe any antitumor activity (ie, time to response and duration of response) of MEDI-538 in this patient population.

Phase 2:

* Determine the overall response in adult patients with CLL who have residual disease following previous therapy for CLL.
* Describe the safety of MEDI-538
* Describe the PK of MEDI-538
* Describe the IM of MEDI-538
* Determine the time to MRD relapse
* Determine the antitumor activity (ie, time to response, duration of response, and time to progression [TTP]) of MEDI-538 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women at least 18 years of age;
* Written informed consent and Heath Insurance Portability and Accountability Act (HIPAA) authorization (applies to covered entities in the USA only) obtained from the patient prior to performing any study-related procedures, including screening visits;
* Previous confirmation of B-cell CLL with a characteristic immunophenotype by flow cytometry;
* MRD positivity, determined by 4-color flow cytometry of bone marrow or peripheral blood in all patients following previous therapy for CLL;
* Measurable and/or residual disease following previous therapy for CLL as follows:

  1. Measurable disease, as determined by NCI-WG criteria, following standard first-line or salvage therapy; this includes patients with PD, SD, or PR (Phase 1 only);
  2. Residual disease as determined by measurable disease (ie, PD, SD, or PR) or by MRD positivity, determined by 4-color flow cytometry of bone marrow and/or peripheral blood in patients with CR or nPR (Phase 2 only);
* Time from completing last therapy for CLL is ≥ 3 months but ≤ 1 year;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
* Presence of live-in companion (relative or friend) who agrees to NOT leave the patient unattended for > 8 hours per day;
* Patient agrees to refrain from engaging in hazardous occupations or activities requiring complete mental alertness such as operating machinery or driving a motor vehicle;
* Females, unless surgically sterile or at least 1 year post-menopausal, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, abstinence, use of a condom with spermicide by the sexual partner or sterile sexual partner) for 21 days prior to the first dose of MEDI-538, and must agree to continue using such precautions through 3 months after the last dose of MEDI-538. Cessation of birth control after this point should be discussed with a responsible physician. Males, unless surgically sterile, must likewise use an effective method of birth control (condom with spermicide) and must agree to continue using such precautions through 3 months after the last dose of MEDI-538;
* Hemoglobin ≥ 10.0 g/dL and platelets > 75.0 x 109/L;
* Total bilirubin ≤ 1.5 x ULN; aspartate transaminase (AST), alanine transaminase (ALT), amylase and lipase ≤ 2 x ULN;
* Serum creatinine ≤ 2 x ULN and creatinine clearance ≥ 50 mL/min;
* Absolute neutrophil count (ANC) > 1.0 × 109/L; and
* For patients who have received previous treatment with alemtuzumab, CD4 counts must be > 200 cells/μL with a negative status for cytomegalovirus (CMV) antigen.

Exclusion Criteria:

* Receipt of MEDI-538 in any previous clinical study;
* History of allergy or reaction to any component of the MEDI-538 formulation;
* History of malignancy other than CLL within 5 years prior to study entry, with the exception of basal cell carcinoma of the skin or carcinoma in situ of the cervix successfully treated with curative therapy;
* Fludarabine-refractory CLL, defined as failure to achieve a PR or CR/nPR to at least one fludarabine-containing regimen, disease progression while on fludarabine treatment, or disease progression in responders within 6 months of last dose of fludarabine;
* Known or suspected CNS involvement;
* Clinical history of significant CNS pathology, eg, uncontrolled headaches, multiple occurrences of confusion, dementia, multiple previous infarcts, or major brain surgery;
* Active infection or known bacteremia. Patients with documented evidence of culture positive sepsis or active infection requiring IV antibiotic therapy must complete a full course of antibiotic treatment with no clinical or laboratory evidence of bacterial infection at least 2 weeks prior to starting therapy with MEDI-538.
* Vaccination (either preventive or therapeutic for infectious disease or cancer) within 2 weeks prior to initiation of MEDI-538;
* Infection with human immunodeficiency virus (HIV-1 or HIV-2), chronic infection with hepatitis B or C, or acute infection with hepatitis A;
* History of serious, chronic autoimmune disease, eg, rheumatoid arthritis, systemic lupus erythematosus, and multiple sclerosis;
* Elective surgery planned during the study period through 30 days after discontinuation of MEDI-538;
* Autologous stem cell transplantation within 26 weeks prior to study entry;
* Allogenic stem cell transplantation or any other solid organ transplant;
* Regular dose of systemic corticosteroids during the 4 weeks prior to initiation of MEDI-538 or anticipated need of corticosteroids exceeding prednisone 20 mg/day or equivalent during the trial, or any other systemic immunosuppressive therapy within 4 weeks prior to study entry;
* Any contraindication to chronic anticoagulation with low-molecular weight heparin (LMWH);
* Inability for safe placement and prolonged use (at least 4 weeks) of a central venous catheter;
* Contraindication to any of the protocol-specified concomitant medications (methylprednisolone, antacids, or antihistamines) during this study;
* Presence of known human anti-murine antibodies or hypersensitivity to immunoglobulins;
* Pregnancy (females of childbearing potential must have a negative urine pregnancy test on the day of the first dose of MEDI-538, prior to dosing) or nursing;
* Evidence of any uncontrolled systemic disease (other than CLL), including autoimmune hemolytic anemia;
* Any finding upon physical examination or history of any disease or behavior that, in the opinion of the investigator or medical monitor, may compromise the safety of the patient in the study or confound the analysis of the study; or
* Inability to meet social environment requirements for outpatient therapy (see Section 3.3.4.2).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-03 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the Phase 1 part of the study are to evaluate the safety, tolerability, and MTD of MEDI-538 by continuous IV infusion for 4 weeks in adult patients with CLL who have measurable disease following previous therapy for CLL. | 30 days after patient's final dose of study drug
The primary objective of the Phase 2 part of the study is to determine the overall response in adult patients with CLL who have residual disease following previous therapy for CLL. | 30 days after patient's final dose of study drug

SECONDARY OUTCOMES:
The secondary outcome of the Phase 1 part of the study include measurement of the PK, IM, and antitumor activity of MEDI-538 in this patient population. | 30 days after patient's final dose of study drug
The secondary objectives of the Phase 2 part of the study include safety, measurement of the PK, IM, and antitumor activity of MEDI-538 in this patient population. | 30 days after patient's final dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kaucic, M.D., Study Director — MedImmune LLC